CLINICAL TRIAL: NCT07363421
Title: Feasibility Study Protocol: TMS-Induced LH Response in Healthy Women in the Luteal Phase
Brief Title: TMS-Induced LH Response in Healthy Women in Luteal Phase
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The City College of New York (Other)
Responsible Party: Principal Investigator, Marom Bikson, Professor, The City College of New York
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2025-0871-CCNY
Record Dates: First submitted 2026-01-21; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Healthy Women
Keywords: LH; FSH; TMS; Blood samples; Hormones

STUDY DESIGN:
Intervention Model Description: This is a single-blind sham controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active (Active Comparator): Transcranial magnetic stimulation of the expected dose will occur
  Interventions: Device: Transcranial Magnetic Stimulation Active
- Sham (Sham Comparator): No transcranial magnetic stimulation of the expected dose will be applied
  Interventions: Device: Transcranial Magnetic Stimulation Sham

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation Active — Participants will receive stimulation to the left DLPFC.
  Stimulation intensity will be standardized based on resting motor threshold.
  Stimulation will be delivered using NeuroStar system.
  Arms: Active
Device: Transcranial Magnetic Stimulation Sham — Participants will undergo identical procedure to the active TMS group, including coil placement, session duration, and acoustic and somatic sensations. A sham device setting will be used that mimics the sound but does not deliver an effective magnetic field to the DLPFC.
  Arms: Sham

SUMMARY:
The purpose of this research is to establish whether non-invasive Transcranial Magnetic Stimulation (TMS), can affect modulation of hormones such: Luteinizing Hormone (LH) and Follicle-stimulating hormone (FSH).

The hypothesis is that applying TMS to the Dorsolateral Prefrontal Cortex with specific pulse patterns, mimicking endogenous Gonodotropin-Releasing Hormone (GnRH) pulses that are known to stimulate LH secretion may modulate hormonal levels.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women aged 22-40 years with regular menstrual cycle.
* In luteal phase at the time of visit.

Exclusion Criteria:

* Presence of any known structural brain abnormalities or tumors.
* Presence of metal implants/devices in the head or neck.
* Has ever had a stroke, seizure, or has a family history of epilepsy.
* Head injury with loss of consciousness.
* Use of hormonal contraceptives in the past 3 months.
* Irregular menstrual cycles.
* Diagnosed with a reproductive system disorder (e.g., PCOS, endometriosis, infertility, hypogonadism).
* History of endocrine disorders such diabetes mellitus, thyroid disease, adrenal disorders, pituitary tumor or others.
* Been diagnosed or received treatment for depression, anxiety disorder, schizophrenia, PTSD or bipolar disorder.
* Have a history of medical disorder such liver or renal impairment, HIV/AIDS or unstable cardiac disease.
* Taking any medications that affect the central nervous system such as antidepressents, antipsychotics, GLP-1 receptor agonists or hormone therapies.
* Are you pregnant, planning pregnancy or breastfeeding.
* Have experienced difficulties in the past during blood draws such as locating the vein, fainting or other adverse reactions.
* Have any sleep disorder such as insomnia or sleep apnea.
* Have fear of needles or the sight of blood.
* Underwent TMS stimulation in the past and had difficulties.

Ages: 22 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Serum luteinizing hormone (LH) and follicle-stimulating hormone (FSH) levels | Six blood draws per participant: Baseline 1 (30 minutes pre-TMS), Baseline 2 (immediately pre-TMS), T1 (20 minutes post-TMS), T2 (55 minutes post-TMS), T3 (20 minutes post-second TMS), T4 (55 minutes pos-second TMS).
  Change in serum LH and FSH concentrations across six time points. Blood samples will be collected via venipuncture. LH and FSH levels will be quantified in IU/L. The primary analysis will evaluate within-subject changes in LH and FSH across the six sampling points and compare hormonal trajectories between active TMS and sham.

SECONDARY OUTCOMES:
Positive and Negative Affect Schedule - Short Form (PANAS-SF) | Baseline and immediately post-intervention
  The PANAS-SF is a self-report questionnaire assessing momentary positive and negative affect. It consists of 20 adjectives (10 positive, 10 negative) rated on a Likert scale (e.g., 1 = very slightly or not at all to 5 = extremely). Separate positive affect and negative affect subscale scores are calculated by summing the relevant items; higher scores indicate greater intensity of that affect dimension.

CONTACTS AND LOCATIONS:
Overall Officials: Marom Bikson, PhD, Principal Investigator — The City College of New York
Locations (1):
- Site 1, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No